CLINICAL TRIAL: NCT06251401
Title: Cardiac Rehabilitation for Breast Cancer Survivors at Risk for Cardiovascular Disease Secondary to Cardiotoxic Treatment
Brief Title: Cardiac Rehabilitation for Breast Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Principal Investigator, Husam Abdel-Qadir, Cardiologist, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-0088-E
Record Dates: First submitted 2024-01-24; First posted 2024-02-09 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer; Cardiovascular Diseases
MeSH Terms: conditions — Breast Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person cardiac rehabilitation (Experimental): Those randomized to in-person cardiac rehabilitation group
  Interventions: Behavioral: In-person supervised cardiac rehabilitation
- Virtual cardiac rehabilitation (Experimental): Those randomized to the virtual, home-based rehabilitation group
  Interventions: Behavioral: Virtual cardiac rehabilitation

INTERVENTIONS:
Behavioral: In-person supervised cardiac rehabilitation — In-person CR consists of weekly group-based supervised exercise training at Women's College Hospital, supplemented with home-based exercise training, with the goal of reaching Canadian Physical Activity Guidelines of 150 minutes a week of moderate-intensity exercise per week. Exercise prescriptions are individualized at baseline by the cardiac rehabilitation team. Both study arms get have the opportunity to attend weekly synchronous virtual group video education sessions for the duration of the 12-week cardiac rehab program with the focus on self-management education and support.
  Arms: In-person cardiac rehabilitation
Behavioral: Virtual cardiac rehabilitation — Virtual CR consists of once-weekly telephone or video conferencing-based follow-ups (according to participant preference and access to internet/smart device) by one of the cardiac rehab providers. Similar to the in-person program, the virtual program also encourages participants to set goals to achieve 150 minutes a week of moderate-intensity exercise. The exercise prescription is individualized to each participant's ability and can vary in number of sessions per week and duration of each exercise session, as per the cardiac rehab provider's discretion. Unlike the in-person program, all these sessions are completed at home in an unsupervised manner. Both study arms get have the opportunity to attend weekly synchronous virtual group video education sessions for the duration of the 12-week cardiac rehab program with the focus on self-management education and support.
  Arms: Virtual cardiac rehabilitation

SUMMARY:
Women with breast cancer treated using anthracyclines and/or trastuzumab are at an increased risk of cardiovascular disease (CVD) following treatment completion. Exercise is known to reduce CVD risk in healthy and several clinical populations, but, whether existing cardiac rehabilitation programs can be leveraged to reduce CVD risk in breast cancer survivors is unknown. This study aims to: i) understand the feasibility of virtual versus in-person cardiac rehabilitation in breast cancer survivors; and ii) compare the effect of virtual versus in-person cardiac rehabilitation on cardiovascular function and injury biomarkers, physical fitness, and psychosocial health. 50 breast cancer survivors with increased CVD risk will be recruited and randomized to either the in-person or virtual arm of the cardiac rehabilitation program at Women's College Hospital (WCH). Data will be collected at baseline, following program completion, and 6-months after program completion. The primary outcomes are measures of study feasibility. Other clinically relevant outcomes to be collected include: i) imaging and blood-based biomarkers of cardiovascular function; ii) physical fitness; iii) objective and self-reported physical activity levels; and iv) self-reported measures of psychosocial wellbeing. These findings will be used to inform the design of a larger-scale cardio-oncology trial and will facilitate development of more comprehensive CVD risk management strategies for breast cancer survivors at WCH.

DETAILED DESCRIPTION:
Rationale Our overarching goal is to support the development of innovative and scalable approaches to CVD prevention in early breast cancer (EBC) survivors. Cardiac rehabilitation (CR) is a cornerstone of both primary and secondary CVD risk management and may be similarly beneficial for survivors at risk of cancer-related CVD. However, it remains unknown if CR-based interventions can reduce CVD risk in those who have received cardiotoxic therapies. Further, the impact of exercise setting (i.e., in-person versus virtual) on intervention safety, adherence, and efficacy has also not been evaluated in this context. Lastly, whether psychosocial wellbeing affects program participation is also not well understood. Ultimately, our study will provide important pilot and feasibility data to inform future randomized trials in this area. It will also lay the foundation for a prospective cohort study that can evaluate the importance of biomarkers and clinical risk factors in predicting future CVD and will provide data that will help identify individuals who are most likely to benefit from aggressive CVD risk factor management.

Design The proposed study is a pragmatic randomized trial of in-person supervised versus virtually delivered CR in EBC survivors treated with anthracyclines and/or trastuzumab. The investigators will also study the evolution of cardiovascular risk markers in women with breast cancer after completion of potentially cardiotoxic chemotherapy.

Objectives and hypotheses

Our specific objectives and related hypotheses are:

1. Primary objective: Assess the feasibility of conducting an adequately powered randomized trial of supervised versus virtual CR in older women (>50 years) with breast cancer who have been treated with anthracyclines and/or trastuzumab Hypothesis: The trial will demonstrate feasibility via the achievement of pre-determined thresholds for participant recruitment, retention, and intervention adherence to CR protocols.
2. Secondary objectives:

   i. Derive estimates of intervention efficacy on markers of cardiac function and injury, aerobic fitness, non-trial physical activity behaviours (i.e., exercise behaviours beyond what is prescribed as part of CR), and psychosocial wellbeing (anxiety, depression, stress) Hypothesis: Improvements in imaging and serum biomarkers, aerobic fitness, and psychosocial measures will be comparable between the two intervention groups.

   ii. Describe the prevalence of abnormal biomarkers from blood, cardiac imaging and stress testing with cardiovascular risk after breast cancer treatment Hypothesis: A substantial proportion of participants will have abnormal global longitudinal strain and serum biomarkers despite having normal LVEF. Estimated aerobic capacity will also be compromised when compared with age- and sex-norms.
3. Tertiary objectives:

   i. Inform the development a novel pathway for cardiometabolic risk reduction for women with breast cancer at WCH, with these data being used to guide out-of-institution scalability Hypothesis: The investigators will identify potential barriers to referral and participation to inform the future development of this program pathway and will be able to determine any cancer-specific needs that may need to be addressed via the program.

   ii. Quantify the differences in intervention delivery costs between the two study arms.

   Hypothesis: Both in-person and virtual CR will be comparable in terms of utilization of consumable resources. Virtual rehabilitation will incur a greater healthcare professional (HCP) time cost for delivery when compared with in-person CR.

   Intervention Briefly, in-person CR consists of once-weekly (or twice weekly if the participant is classified is being high risk, i.e., elevated blood pressure with exercise, or <85% age-predicted aerobic fitness) group-based supervised exercise training at WCH, supplemented with home-based exercise training, with the goal of reaching Canadian Physical Activity Guidelines of 150 minutes a week of moderate-intensity exercise per week. Exercise prescriptions are individualized at baseline by the CR team based on a symptom-limited stress test. Virtual CR consists of once-weekly telephone or video conferencing-based follow-ups (according to participant preference and access to internet/smart device) by one of the HCPs. Similar to the in-person program, the virtual program also encourages participants to set goals to achieve 150 minutes a week of moderate-intensity exercise. The exercise prescription is individualized to each participant's ability and can vary in number of sessions per week and duration of each exercise session, as per the HCP's discretion. Unlike the in-person program, all these sessions are completed at home in an unsupervised manner. Additionally, both study arms get have the opportunity to attend weekly synchronous virtual group video education sessions for the duration of the 12-week CR program with the focus on self-management education and support. The program's Registered Dietitian, Social Worker, and Pharmacist (who teach some of the education sessions) may offer 1:1 visits with the participants if necessary.

   Statistical Analysis Participant demographics, clinical characteristics (including prevalence of abnormal biomarkers), and feasibility metrics (including reasons for non-participation) will be analyzed using descriptive statistics (mean ± standard deviation, and frequency (%), as applicable). Exercise and education session attendance will be reported as the proportion attended and compared between groups using the chi-square test (or Fisher's exact test, as appropriate). Exercise prescription adherence will be reported as the average percentage of exercise completed relative to exercise dose prescribed and will be compared between groups using independent-samples t-tests (or Wilcoxon Rank Sum test, as appropriate).

ELIGIBILITY:
Inclusion Criteria:

* age > 50 years
* previous receipt of anthracyclines and/or trastuzumab for breast cancer
* ability to participate in in-person cardiac rehabilitation

Exclusion Criteria:

* medical contraindications that preclude safe exercise participation17
* unwillingness to comply with study protocols.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 1 week after study completion
  Defined as number of patients who agree to participate relative to the number of patients approached.
Intervention safety | 1 week post-intervention
  Data on all intervention-related adverse events (as defined by the Common Terminology Criteria for Adverse Events [CTCAE]) will be collected and reported according to CTCAE-defined categories. Non-trial related adverse events during the intervention period will also be recorded given that they may significantly impact participation.
Study retention | 1 week post-intervention
  Retention will be assessed by measuring attrition throughout the intervention period.
Reasons for drop-out | 1 week post-intervention
  Reasons for dropout and/or non-compliance to assessment protocols will also be collected.
Intervention adherence | 1 week post-intervention
  Exercise adherence will be collected as relative dose intensity (RDI; exercise dose performed in each session relative to prescribed exercise dose).
Participant satisfaction | 1 week post-intervention
  Satisfaction with the intervention and participant experiences will be collected via an investigator-created survey.

SECONDARY OUTCOMES:
Estimated aerobic fitness | 2 weeks before starting cardiac rehabilitation and 1 week after completing cardiac rehabilitation
  Estimated peak aerobic fitness using a prediction equation and symptom-limited stress test, using either the Bruce or modified Bruce protocol completed prior to the first cardiac rehab exercise session and at program completion.
Left ventricular ejection fraction (LVEF) | 2 weeks before starting cardiac rehabilitation, 1 week after completing cardiac rehabilitation, and 6 months after completing cardiac rehabilitation
  Volumetric determination of LVEF assessed via electrocardiography in accordance with practice guidelines.
Global longitudinal strain (GLS) | 2 weeks before starting cardiac rehabilitation, 1 week after completing cardiac rehabilitation, and 6 months after completing cardiac rehabilitation
  Determination of GLS via strain analysis assessed using electrocardiography
E/A ratio | 2 weeks before starting cardiac rehabilitation, 1 week after completing cardiac rehabilitation, and 6 months after completing cardiac rehabilitation
  Measure of diastolic dysfunction assessed via electrocardiography in accordance with practice guidelines.
Duke Activity Status Index | 2 weeks before starting cardiac rehabilitation, 1 week after completing cardiac rehabilitation, and 6 months after completing cardiac rehabilitation
  Self-reported measure of physical activity
Godin Leisure Time Exercise Questionnaire | 2 weeks before starting cardiac rehabilitation, 1 week after completing cardiac rehabilitation, and 6 months after completing cardiac rehabilitation
  Self-reported measure of physical activity
Beck Depression Inventory | 2 weeks before starting cardiac rehabilitation, 1 week after completing cardiac rehabilitation, and 6 months after completing cardiac rehabilitation
  Self-reported assessment of depression
Short-form survey (SF-36) | 2 weeks before starting cardiac rehabilitation, 1 week after completing cardiac rehabilitation, and 6 months after completing cardiac rehabilitation
  Self-reported measure of quality of life
Work Limitations Questionnaire | 2 weeks before starting cardiac rehabilitation, 1 week after completing cardiac rehabilitation, and 6 months after completing cardiac rehabilitation
  Self-reported assessment of degree to which individual's condition affects ability to return to work
Automated Self-Administered Dietary Assessment Tool (ASA24) | 2 weeks before starting cardiac rehabilitation, 1 week after completing cardiac rehabilitation, and 6 months after completing cardiac rehabilitation
  Self-reported measure assessing individual's diet
Objective assessment of physical activity levels | 1 week after completing cardiac rehabilitation
  Participants will be provided Fitbits for the duration of their participation in cardiac rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Husam Abdel-Qadir, MD-PhD, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada